CLINICAL TRIAL: NCT05813158
Title: Comparing the Perioperative Analgesic Effect of Two Different Volumes of Local Anesthetic Solution in Erector Spinae Plane Block in Patients Undergoing Modified Radical Mastectomy A Randomized Comparative Study
Brief Title: Comparing the Perioperative Analgesic Effect of Two Different Volumes of Local Anesthetic Solution in Erector Spinae Plane Block in Patients Undergoing Modified Radical Mastectomy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Yasmina sayed Abdrabo Ismael (Unknown); Norhan Abdelaleem Ali (Unknown); Ahmed Shaker Ragab (Unknown)
Responsible Party: Principal Investigator, Ahmed Abdalla, Professor of Anesthesia &I.C.U and Pain Clinic, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: N-44-2022/MSc
Record Dates: First submitted 2022-11-18; First posted 2023-04-14 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Comparing of 2 Different Volumes in ESPB in Patients Undergoing MRM

STUDY DESIGN:
Intervention Model Description: We hypothesize that high volume low concentration ultrasound-guided Erector Spinae Plane block is going to be more effective than low volume high concentration in patients undergoing MRM. Many authors advocate increasing the volume of injection in fascial plane blocks to allow better spread of local anesthetic according to multiple studies
Who Masked: Participant, Investigator
Masking Description: Patients will be randomly allocated to one of the two groups by sealed closed envelop technique
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Patients will preoperatively receive low concentration-high volume U/S ESP block, and then the patient will be transferred to the operating room one syringe of 30ml bupivacaine 0.25% {15 ml bupivacaine 0.5% and 15ml normal saline}, for each patient.
  Interventions: Drug: Group 1(low concentration-high volume bupivacaine US guided Erector Spinae Plane block)
- Group 2 (Active Comparator): Patients will preoperatively receive high concentration-low volume U/S ESP block block, and then the patient will be transferred to the operating room one syringe of 15 ml bupivacaine 0.5% {15 ml bupivacaine 0.5% }, for each patien).
  Interventions: Drug: Group 2(high concentration-low volumecbupivacaine US guided Erector Spinae Plane block)

INTERVENTIONS:
Drug: Group 1(low concentration-high volume bupivacaine US guided Erector Spinae Plane block) — Patients will preoperatively receive low concentration-high volume ultasound guided Erector Spinae Plane block, and then the patient will be transferred to the operating room ) one syringe of 30ml bupivacaine 0.25% {15 ml bupivacaine 0.5% and 15ml normal saline} for each patient
  Other Names: Erector Spinae Plane Block with high volume-low concentration bupivacaine 0.25%
  Arms: Group 1
Drug: Group 2(high concentration-low volumecbupivacaine US guided Erector Spinae Plane block) — Patients will preoperatively receive high concentration-low volume ultasound guided Erector Spinae Plane block, and then the patient will be transferred to the operating room (one syringe of 15 ml bupivacaine 0.5% {15 ml bupivacaine 0.5% } for each patien).
  Other Names: Erector Spinae Plane Block with low volume-high concentration bupivacaine 0.25%
  Arms: Group 2

SUMMARY:
The aim of this study is to compare and evaluate the analgesic effects of ultrasound-guided Erector Spinae Plane block using low volumes and high concentrations versus high volumes and low concentrations in patients undergoing MRM.

DETAILED DESCRIPTION:
Multiple regional techniques have been developed in recent years for postoperative analgesia of breast surgery including ESPB aiming to be effective and associated with less complications when compared to the gold standard techniques (thoracic epidural analgesia or paravertebral block)..

Ultrasound guided erector spinae plane (ESPB) block was described in 2016 as a novel regional anesthetic technique for acute and chronic thoracic pain, it has been used as a regional anesthetic technique for breast surgery based on case reports and case series. It is a paraspinal fascial plane block that involves injection of local anesthetic deep in the erector spinae muscle and superficial to the tips of the thoracic transverse processes. The site of injection is distant from the pleura, major blood vessels, and spinal cord; hence, performing the ESPB has relatively few contraindications. The injected local anesthetic drug blocks the ventral and dorsal rami of spinal nerves on the paravertebral area .

Multiple studies have reported improved efficiency of interfascial blocks by increasing the volume of injection promoting better spread of local anesthesia. According to the authors best knowledge there is no studies comparing different volumes and concentration in ESPB in patients undergoing MRM This study aims to see the effect of fixing the drug mass of anaesthetic given in both groups, while altering the concentration of the anesthetic and total volume administered. One group will receive a lower concentration and higher volume, while the other will receive a higher concentration and lower volume.

ELIGIBILITY:
Inclusion Criteria:

Age starting from 18 to 60 years.

* Genders eligible for study: female sex.
* ASA II-III.
* Patients undergoing modified radical mastectomy.
* Body mass index (BMI) from 18.5 to 30 kg/m2.

Exclusion Criteria:

Patient refusal

* Known allergy to local anesthetics
* Bleeding disorders; platelets count <50,000, prothrombin concentration <60% or any coagulopathy disorder.
* Use of any anti-coagulants
* Inability to provide informed consent
* ASA IV
* Neurological disorders
* Patient with psychiatric disorders

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Total dose of morphine needed postoperatively | Through Study Completion Up to 1 Day
  Total dose of morphine needed postoperatively

SECONDARY OUTCOMES:
Time to first rescue analgesia, starting after extubation | Through Study Completion over the first 24 hours postoperative
  Time to first rescue analgesia, starting after extubation
Duration of surgery | Through Study Completion 24 hours postoperative
  Duration of surgery
Blood loss, | Through Study Completion,an average of 1day
  Blood loss,
Total dose of fentanyl required intraoperative (including induction dose) | Through study completion,an average of 1day
  Total dose of fentanyl required intraoperative (including induction dose)
Pain score at 15, 30, 45 and 60 min., 3,6,12 and 24 h after surgery | through study completion,an average of 1day
  Pain score at 15, 30, 45 and 60 min., 3,6,12 and 24 h after surgery
Need for blood transfusion | Through Study Completion over the first 24 hours postoperative
  Need for blood transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abdalla Mohamed, M.D, Principal Investigator — Cairo University
Locations (1):
- Ahmed Abdalla Mohamed, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Till Study Ending